CLINICAL TRIAL: NCT04640662
Title: The Effects of Platelet Rich Plasma Versus Prolotherapy on Pain and Function in Rotator Cuff Tendinopathy: A Randomized Clinical Trial
Brief Title: The Effects of Platelet-Rich Plasma Versus Prolotherapy On Rotator Cuff Tendinopathy: A Randomized Controlled Trial.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Samihah Abdul Karim, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PV062-2018
Record Dates: First submitted 2020-11-11; First posted 2020-11-23 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Rotator Cuff Tendinosis; Supraspinatus Strain; PRP
Keywords: Platelet-rich plasma; Prolotherapy; Biologics; Tendinopathy
MeSH Terms: conditions — Rotator Cuff Injuries; Tendinopathy | interventions — Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-Rich plasma (Experimental): 2 ml PRP using commercial kit- YCell Biokit
  Interventions: Biological: Platelet-Rich Plasma; Biological: Prolotherapy
- Prolotherapy (Active Comparator): 2 ml 16.5% Dextrose solution
  Interventions: Biological: Platelet-Rich Plasma; Biological: Prolotherapy

INTERVENTIONS:
Biological: Platelet-Rich Plasma — Single-injection of 2 ml PRP into the lesion under ultrasound-guided
  Other Names: PRP
Biological: Prolotherapy — Single-injection of 2ml dextrose 16.5% into the lesion under ultrasound-guided
  Other Names: Prolo

SUMMARY:
Rotator cuff tendinopathy is the common cause of shoulder pain in the working-age group and the elderly (1). The condition reported takes an average of 10 months or longer to recover. Treatment ranges from non-surgical therapy through exercise, physiotherapy, injections to surgery (2). Injection of steroid was used in many cases to reduce pain. However, steroid only provided short term pain relief and did not resolve the main pathology. Emerging of biologics agents such as platelet-rich plasma (PRP) and prolotherapy are alternative to the treatment (3). PRP is a concentrated platelet which contains a high concentration of protein that helps in the healing process (4). Prolotherapy with the commonly used substance dextrose works by attracting inflammatory substrate and stimulate own body healing process (5).

This study takes place at the University of Malaya Medical Centre. Participants diagnosed with rotator cuff tendinopathy are randomly divided into two groups- Platelet Rich Plasma (PRP) group and Prolotherapy group. All participants are screened by the researcher for the eligibility to join the study. Subsequently, the participants undergo baseline assessment on the clinical, functional, biomechanics and ultrasound. Blood is taken in all patient, to make the patient blind to the intervention they received. In the PRP group- the participants received 2ml of PRP, and in prolotherapy group, the participants received 2ml of 16.5% dextrose solution. A single injection is done by an experienced Sports Physician using ultrasound-guided into the injured area. The assessor at baseline, and follow up are blinded to the intervention. The participants need to come for follow up at 3 weeks, 6 weeks, 3 months and 6 months after injection.

Systematic reviews showed the benefit of biologics agent to treat tendon injuries, especially for lateral epicondylitis and patellar tendinitis (6). Many studies for soft tissue injury were on PRP compared to prolotherapy. This study hypothesized that both treatments result in significant improvement in pain and function after the intervention. PRP might provide more significant improvement compared to prolotherapy.

DETAILED DESCRIPTION:
Study design This study is a randomized, double-blind, controlled trial conducted at the University of Malaya Medical Centre, Kuala Lumpur, Malaysia.

Patients The patients will be recruited from the following clinics: Sports Medicine, orthopaedic, rheumatology, outpatient and staff health. Notice of study invitation in this study will be distributed to all the respective clinic. Patients with a confirm diagnosis of supraspinatus tendinopathy by ultrasound or MRI will be invited to participate in this study. Study screening will be carried out to ensure the inclusion and exclusion criteria are fulfilled by the research team in Sports Medicine Clinic.

Procedures

PRP group Patients under PRP group will receive a single 2 mL injection of PRP into the injury site under ultrasound guidance administered by a sports physician. The PRP will be prepared using a commercial kit, Y-Cell BioKit Systems.

Prolotherapy group Patients in the prolotherapy group will receive a single 2 mL injection of 16.5% dextrose solution administered under ultrasound guidance.

Injection technique Injection will be performed in the Sports Medicine Clinic using aseptic technique. Both the PRP and prolotherapy will be prepared in a syringe and covered with a black tape to ensure the patients did not know the content of the syringe. Patients will be placed in the supine position and will be requested not to turn their head during the procedure. A 22 G needle will be used for injection under ultrasound guided.

Following injection, cryotherapy will be applied for 15 min. Upon discharge, patients will be advised to rest the injected shoulder for the next 48 hours and to avoid taking NSAIDs.

Rehabilitation program Patients will receive a booklet for shoulder stretching and strengthening exercise. A logbook will be provided for the patients to record their exercise session. Rehabilitation sessions will be advise to commenced only day three of injection.

Sample size The sample size was estimated based on the primary outcome of functional score. Improvement was defined by a decrease in the mean Shoulder Pain and Disability Index (SPADI) of 17.7 ± 3.7 in the platelet-rich plasma group11 and 16.12 ± 12.8211 for prolotherapy. For this study, the sample size was calculated after taking into account the desired statistical significance level set at 5%, and the power of the study set at 80%, with type I error rate of less than 0.05 is permitted and a false-negative rate of less than 0.20. The sample size is calculated using the G*Power version 3.1.9.2 software11. With the assumption of 30% drop out, hence, to detect a difference in the functional outcome, a minimum of 30 patients in each group is required.

Randomization Randomization will be performed using computer-generated block randomization of ten. Subjects will be randomized into either PRP group or Prolo group.

Blinding The patients and assessors will be blind to the intervention. Two sports physician who not directly involved in the randomization and injection will perform the outcome measure assessment.

Outcomes

Patients characteristics Patients sociodemographic information, including gender, date of birth, ethnic background, job description and recreational activities will be recorded. Information related to the shoulder pain such as duration and other past rehabilitation and treatment will also be documented.

Primary outcome measures The primary outcome of this study is pain score using the visual analog score (VAS) score and shoulder function using shoulder pain and disability index (SPADI) score.

VAS score (7) is a continuous scale, 10 cm length with the left most anchor indicate "no pain" (0) to "extreme pain" (10).

SPADI was used to measure shoulder pain and disability in an outpatient setting within the recent 1 week. It contains 13 items that assess pain and disability. SPADI reveals good construct validity, correlating well with other specific shoulder questionnaires and responsive to change over time (8).

Secondary outcome measures

1. Constant-Murley score assessed four aspects of shoulder injury which consist of two subjective item- pain and activities of daily living (ADL) and two objective item- range of motion (ROM) and strength. This score was used in many shoulder studies and had good response to change quality (9).
2. Clinical test which consist of special test
3. Biomedical test which consist of shoulder ROM using goniometer, strength using dynamometer and periscapular muscle activities using electromyogram.
4. Adverse effect of the injections will also be recorded.

Data collection and management Data will be collected from patients at baseline, 3 weeks, 6 weeks, 3 months and 6 months. All data collected will be stored securely in a locked cabinet in Sports Medicine Department throughout the trial and only can be access by the researcher involved. To ensure confidentiality, each patient will have the trial identification number.

Statistical analysis The outcome variables will be analyzed with the principle of intention-to-treat (ITT). The mean VAS score and SPADI between groups will be compared using either the parametric independent t-test or non-parametric test using Mann-Whitney U test. The secondary outcome measures will be examine using linear mixed- model analysis. All statistical analysis will be performed using the SPSS V.25.0 (SPSS), and a p value of <0.05 will be considered to be significant.

Ethics and dissemination The study was approved by the Medical Research Ethics Committee of the University of Malaya Medical Centre (MREC ID: 201977-7623). This trial was registered at the National Medical Research Register (NMRR-19-1658-48279). Participation in this study is strictly voluntary. Possible patients will be informed of all the procedures involved in the reserach verbally and by the patient's information sheets. Patients will be required to sign the informed consent form before participation. Patient will be allowed to withdraw from the study at any time. Results from this study will be presented at scientific conferences and publish in journal.

ELIGIBILITY:
Inclusion Criteria:

* Chronic shoulder pain more than 3 months
* Diagnosis of supraspinatus tendinopathy by Sports Physician or Orthopaedic
* Diagnosis by ultrasound or MRI

Exclusion Criteria:

* Patients with the following medical condition: autoimmune rheumatology disease, blood disorder
* Patients with the following shoulder conditions: referred pain from cervical, recent shoulder surgery, shoulder instability, complete rotator cuff tear, adhesive capsulitis
* Patients with the following medications: anti-coagulant treatment, steroid injection in less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Pain Reduction change from baseline | 3 weeks, 6 weeks, 3 months and 6 months
  Visual analog score (VAS) score will be used. The scale is between 0 to 10; 0 is no pain, 10 is the worst pain imaginable
Functional score change from baseline | 3 weeks, 6 weeks, 3 months and 6 months
  Shoulder Pain and Disability Index (SPADI) questionnaire Two subscales namely pain and disability. Pain scale is from 0 to 10; 0 is no pain, 10 is the worst pain imaginable
  Disability scale range from 0 to 10; 0 no difficulty, 10 is so difficult it requires help

SECONDARY OUTCOMES:
Strength in kg | 3 weeks, 6 weeks, 3 months and 6 months
  The test will use Commander Dynamometer. The changes in strength (kg) from baseline will be assessed during each follow up
Range of Movement | 3 weeks, 6 weeks, 3 months and 6 months
  Goniometer will be used for the assessment. The changes in the range of motion in degrees from baseline will be assessed at all follow up
Peri-scapular Muscle activity | 6 weeks, 3 months and 6 months
  Electromyogram will be used for the assessment. Muscle amplitude will be recorded at baseline and at follow up
Ultrasound findings The parameters will be on tendon thickness, neo-vascularaization and tear size | 6 weeks, 3 months and 6 months
  The ultrasound of the supraspinatus will be assessed to look for changes in the tendinopathy characteristics at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Samihah A. Karim, MD, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Centre, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing for the following:
  * Study Protocol
  * Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after completion in September 2021 to 2025
Access Criteria: The IPD will be shared with a fellow researcher who interested with the topic. Analysis for systematic review such as the study protocol and the result will be shared through open assess or upon request.

REFERENCES:
- [Background] Lin MT, Chiang CF, Wu CH, Huang YT, Tu YK, Wang TG. Comparative Effectiveness of Injection Therapies in Rotator Cuff Tendinopathy: A Systematic Review, Pairwise and Network Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2019 Feb;100(2):336-349.e15. doi: 10.1016/j.apmr.2018.06.028. Epub 2018 Aug 2. PMID 30076801
- [Result] 1. Littlewood, C., S. May, and S. Walters, Epidemiology of Rotator Cuff Tendinopathy: A Systematic Review. Shoulder & Elbow, 2013. 5(4): p. 256-265.
- [Result] Lewis J, McCreesh K, Roy JS, Ginn K. Rotator Cuff Tendinopathy: Navigating the Diagnosis-Management Conundrum. J Orthop Sports Phys Ther. 2015 Nov;45(11):923-37. doi: 10.2519/jospt.2015.5941. Epub 2015 Sep 21. PMID 26390274
- [Result] Hurley ET, Hannon CP, Pauzenberger L, Fat DL, Moran CJ, Mullett H. Nonoperative Treatment of Rotator Cuff Disease With Platelet-Rich Plasma: A Systematic Review of Randomized Controlled Trials. Arthroscopy. 2019 May;35(5):1584-1591. doi: 10.1016/j.arthro.2018.10.115. Epub 2019 Apr 15. PMID 31000394
- [Result] Trebinjac S and Kitchbi. Long-term effect of Prolotherapy on symptomatic rotator cuff tendinopathy. Journal of Health Sciences 2015;5(3):93-98
- [Result] Docheva D, Muller SA, Majewski M, Evans CH. Biologics for tendon repair. Adv Drug Deliv Rev. 2015 Apr;84:222-39. doi: 10.1016/j.addr.2014.11.015. Epub 2014 Nov 21. PMID 25446135

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04640662/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT04640662/ICF_000.pdf